CLINICAL TRIAL: NCT00357526
Title: YOUNG WOMEN'S EXPERIENCES: ORAL CONTRACEPTIVE PILLS VS The VAGINAL RING
Brief Title: Oral Contraceptive Pills Compared to Vaginal Rings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Organon (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H10857-19674-04
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2006-03

CONDITIONS: Pregnancy
Keywords: vaginal ring; Oral contraceptive pills; Teenagers; Young women; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Contraceptive Devices, Female

INTERVENTIONS:
Drug: OCPs
Device: vaginal ring

SUMMARY:
The purpose of this study is to determine whether teens and young women would prefer the Nuvaring to oral contraceptive pills after having tried both methods.

DETAILED DESCRIPTION:
Sexually active young women (n=130), aged 15-21 years, were randomly assigned to use either the vaginal ring or oral contraceptive pills for an initial study interval of three 28-day cycles, followed by three cycles of the alternate method. Participants completed surveys about method use, acceptability and side effects at baseline, after three cycles, and after six cycles, as well as in a follow up telephone interview one month after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active young women (n=130), English or Spanish speaking, aged 15-21 years, able and willing to try oral contraceptives and vaginal rings for 6 months

Exclusion Criteria:

* Not able or willing to use hormonal contraceptives, moving out of the area, pregnant or intending to become pregnant during the study time frame, not sexually active

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130
Dates: Start 2003-04; Study Completion 2004-08

PRIMARY OUTCOMES:
Satisfaction

SECONDARY OUTCOMES:
Compliance
Acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Stewart, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- New Generation Health Center, San Francisco, California, United States